CLINICAL TRIAL: NCT06749158
Title: Radiographic and Histological Assessment of Guided Bone Regeneration Using Deproteinized Bovine Bone Compared to Spontaneous Bone Regeneration of Maxillary Defects , Resulted from Enucleation of Intra-bony Cystic Lesions : Randomized Control Clinical Trial
Brief Title: Radiographic and Histological Assessment of GBR Using DBB Compared to Spontaneous Bone Regeneration of Maxillary Defects , Resulted from Enucleation of Intra-bony Cystic Lesions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Mohamed Abdelzaher, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBO-CU.2024
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-10

CONDITIONS: Maxillary Cyst
Keywords: Guided bone regeneration; Spontaneous bone regeneration

STUDY DESIGN:
Who Masked: Participant
Masking Description: This trial is considered a randomized single blind clinical trial due to the following:
  * The participants will be blinded to the technique that will be used during the surgical procedure.
  * The operator will not be blinded for both techniques during the surgical procedure as the two techniques are different.
  * The outcome assessor cannot be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- spontaneous bone regeneration (Active Comparator): after cyst enucleation, the intra-bony defect will be covered by Titanium mesh that is fixed by mono-cortical titanium screws.
  Interventions: Procedure: spontaneous bone regeneration
- guided bone regeneration (Experimental): cyst enucleation will be followed by filling the intra-bony defect with Deproteinized Bovine Bone.
  -Titanium mesh will cover the bone window completely and will be fixed to the bone using mono-cortical titanium screws.
  Interventions: Procedure: guided bone regeneration

INTERVENTIONS:
Procedure: spontaneous bone regeneration — stage 1 surgery:
  1. after administration of Local anesthesia (articaine hydrochloride 68 mg/1.7 ml + adrenaline 0.017 mg/1.7 ml injectable solution), sulcular incision will be done , extending two teeth beyond the area of interest followed by two oblique incisions on either side of the flap
  2. after flap elevation, enucleation of the cystic lesion and extraction of the non-restorable teeth related to the lesion will be done.
  3. titanium mesh will be tailored with 3 mm overlap at the edges to cover the bone window completely and fixed to the bone using mono-cortical titanium screws.
  This will be followed by:
  * proper decompression of soft tissue to achieve tension-reduced suture.
  * Primary closure will be performed using 4-0 vicryl sutures.
  * Sutures will be removed one week postoperatively. stage 2 surgery(after 6 months):
    1. titanium mesh and screws will be removed.
    2. core biopsy will be obtained for histological assessment
    3. implant/s placement.
  Arms: spontaneous bone regeneration
Procedure: guided bone regeneration — stage 1 surgery after cyst enucleation and extraction of the non-restorable teeth related to the lesion, The intra-bony defect will be filled with Deproteinized Bovine Bone.
  * Titanium mesh will be tailored with 3mm overlap at the edges to cover the bone window completely and fixed to the bone using mono-cortical titanium screws. This will be followed by:
  * proper decompression of soft tissue will be applied to achieve tension-reduced suture.
  * Primary closure will be performed using 4-0 vicryl sutures.
  * Sutures will be removed one week postoperatively. stage 2 surgery(6 months later) :
    1. titanium mesh will be removed.
    2. core biopsy will be obtained for histological assessment.
    3. implant/s placement.
  Arms: guided bone regeneration

SUMMARY:
Two groups of patients with maxillary defects resulted from enucleation of intra-bony cystic lesions One will be subjected to guided bone regeneration while the other group will be subjected to spontaneous bone regeneration.

DETAILED DESCRIPTION:
* Two groups of patients with maxillary cystic lesions indicated for enucleation. One will be subjected to guided bone regeneration while the other will be subjected to spontaneous bone regeneration.
* General pre-operative procedures:

  * All patients will undergo appropriate preparation involving periodontal therapy , proper oral hygiene measures in addition to endodontic treatment for the non-vital teeth related to the lesion.

intraoperative procedure: (both groups)

* Scrubbing and draping of the patient will be carried out in a standard fashion using betadine surgical scrub.
* Local anesthesia will be administered (articaine hydrochloride 68 mg/1.7 ml + adrenaline 0.017 mg/1.7 ml injectable solution.
* Flap design: a sulcular incision will be done , extending two teeth beyond the area of interest followed by two oblique incisions on either side of the flap. A full thickness mucoperiosteal flap will be raised to expose the area occupied by the lesion.
* After flap reflection, the exposed bone related to the lesion will need to be removed to provide adequate accessibility before enucleation of the lesion.
* The specimens will be fixed in 10% formalin for pathological examination.

Intra-operative procedures - continued in Study Group (GBR group) The intra-bony defect will be filled with Deproteinized Bovine Bone. In Both groups: Titanium mesh will be tailored with 3mm overlap at the edges to cover the bone window completely and fixed to the bone using mono-cortical titanium screws.

This is followed by:

* proper decompression of soft tissue will be applied to achieve tension-reduced suture.
* Primary closure will be performed using 4-0 vicryl sutures.
* Sutures will be removed one week postoperatively.

Postoperative medications:

For both groups, postoperative antibiotic course of amoxicillin+ clavulanic acid 1 g tab (Augmentin) will be prescribed for one week and isobutylphenylpropionic acid 600 mg tab (Brufen) twice daily for one week. One shot of dexamethasone 8 mg vial will be administered intramuscularly immediately after the surgery together with ketorolac tromethamine 30 mg .

Postoperative care and instructions:

* Cold compresses will be applied for 10 minutes every 30 minutes for the first 24 hours postoperatively replaced by warm fomentation with the same rate for the next two days.
* Patients will be advised to maintain good oral hygiene and oral hygiene rinses using 2% chlorohexidine gluconate mouth rinse for a week starting from the second postoperative day (three times daily)
* Soft diet is recommended for the first 48 hours.
* The patients will be recalled after two days, after one week, at the end of the first month and then at three and six months to monitor the soft tissue healing where the sutures were removed after one week, then at the sixth months to evaluate the bony healing.

Radiographic assessment will be achieved by CBCT scan immediately postoperative to determine the baseline bone density and 6 months postoperatively to evaluate the change in the bone density . A total of three scans will be taken for each patient.

6 months after the surgery ,titanium mesh and the screws will be removed , core biopsy will be taken for histological assessment and implant/s will be placed.

ELIGIBILITY:
Inclusion Criteria:

* Pathological Maxillary intra-bony defects with diameter ranging from 1.5 to 4.0 cm.
* patients indicated for implant placement after teeth extraction.
* Age range from 20-50 years.
* Patients free from any systemic conditions and bone metabolism diseases that might interfere with the surgical intervention, soft tissue or hard tissue healing.
* No evidence of acute inflammation.
* Regular attendance at control visits.

Exclusion Criteria:

* Pregnancy or lactation.
* Systemic conditions that compromise bone healing such as : uncontrolled diabetes mellitus, history of chemotherapy or radiotherapy or Hematological disorders.
* Patients taking bisphosphonates, glucocorticoids or other drugs that may interfere with bone metabolism.
* presence of infection at the surgical site.
* infected cysts and odontogenic keratocyst.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
The amount of change in the Bone density | 6 months postoperatively
  Measuring the amount of change in the bone density using cone beam computed tomography in hounsfield unit

SECONDARY OUTCOMES:
Percentage of bone area | 6 months postoperatively
  Measuring the percentage of bone area using Histomorphometric analysis of decalcified bone sections with hematoxylin and eosin(H&E) stain using image analyzer computer system.

OTHER OUTCOMES:
Percentage of mature bone | 6 months postoperatively
  Measuring the percentage of mature bone using Histomorphometric analysis of decalcified bone sections with Masson's trichrome stain using image analyzer computer system.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Abdelrasoul, PhD, Study Director — faculty of oral and dental medicine, Cairo university
Locations (1):
- faculty of oral and dental medicine, Cairo university, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Radiographic bone volume alteration after jaw cyst enucleation with or without simultaneous bone grafts: A prospective randomized study — https://pubmed.ncbi.nlm.nih.gov/35576245/
- See also: Review Int J Oral Sci . 2020 Dec 30;12(1):37. doi: 10.1038/s41368-020-00107-z. Titanium mesh for bone augmentation in oral implantology: current application and progress — https://pubmed.ncbi.nlm.nih.gov/33380722/
- See also: Jaw cysts - filling or no filling after enucleation? A review — https://pubmed.ncbi.nlm.nih.gov/21890372/
- See also: Bone Grafts and Substitutes in Dentistry: A Review of Current Trends and Developments — https://pubmed.ncbi.nlm.nih.gov/34070157/
- See also: Barrier Membranes for Guided Bone Regeneration (GBR): A Focus on Recent Advances in Collagen Membranes — https://pubmed.ncbi.nlm.nih.gov/36499315/